CLINICAL TRIAL: NCT00126412
Title: An Open-Label, Multicentre, Phase 3 Scintigraphy Study Assessing 123I-mIBG Uptake in Subjects Being Evaluated for Phaeochromocytoma or Neuroblastoma
Brief Title: Meta-Iodobenzylguanidine (123I mIBG) Scintigraphy in Patients Being Evaluated for Phaeochromocytoma or Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MBG308
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Pheochromocytoma; Neuroblastoma
Keywords: Phaeochromocytoma; Neuroblastoma; diagnosis; 123I-mIBG
MeSH Terms: conditions — Pheochromocytoma; Neuroblastoma; Disease | interventions — 3-Iodobenzylguanidine

ARMS (1):
- 123I-mIBG (Meta-iobenzylguanidine) (Experimental): All subjects received 123I-mIBG injection over at least 1 to 2 minutes through a cannula (or indwelling catheter in the vein). After the injection of 123I-mIBG was complete, the cannula was flushed with at least 5 mL of 0.9% sodium chloride solution over a maximum of 10 seconds.
  All subjects ≥18 years of age and children with a weight of ≥70 kg were to receive an intravenous injection of 370 ±10% MBq (333 to 407 MBq [9.0 to 11 mCi] of 123I-mIBG). Doses of 123I-mIBG for children <18 years of age (with a weight of 8-70 kg) were to be calculated on the basis of a reference activity for an adult scaled to body weight according to the schedule proposed by the European Association of Nuclear Medicine (EANM) Paediatric Task Group; for children <8 kg, a scaled activity or a fixed minimum activity of 80 ±10% MBq (72 to 88 MBq [1.9 to 2.2 mCi]) was permissible.
  Interventions: Drug: 123I-mIBG (meta-iodobenzylguanidine)

INTERVENTIONS:
Drug: 123I-mIBG (meta-iodobenzylguanidine)
  Other Names: Iobenguane; mIBG

SUMMARY:
The study is designed to study the effectiveness of 123I-mIBG as a diagnostic imaging agent in evaluating patients with known or suspected neuroblastoma or phaeochromocytoma.

ELIGIBILITY:
Inclusion Criteria:

For subjects recruited under Amendment 01 :

(1) a) The subject has known or suspected neuroblastoma and is undergoing evaluation of disease status (for which a 123I-mIBG scintigraphic examination is clinically appropriate) OR b) The subject is ≥18 years of age with either: i) Known phaeochromocytoma. ii) Suspected phaeochromocytoma based on abnormal levels of catecholamines or metabolites in the urine or blood with difficult to control chronic or paroxysmal hypertension and/or abnormalities in the adrenal region on ultrasound, computerised tomography (CT), or magnetic resonance imaging (MRI). iii) A diagnosis of a familial or hereditary condition known to be associated with phaeochromocytoma (multiple endocrine neoplasia, von Hippel-Landau disease, neurofibromatosis, etc).

For subjects recruited under Amendment 02 :

1. a) The subject has known or suspected neuroblastoma and is undergoing evaluation of disease status (for which a 123I-mIBG scintigraphic examination is clinically appropriate) OR b) The subject has either: i) Known phaeochromocytoma, or, ii) Suspected phaeochromocytoma based on abnormal levels of catecholamines or metabolites in the urine or blood in conjunction with difficult to control chronic or paroxysmal hypertension and/or abnormalities in the adrenal region on ultrasound, CT, or MRI, or iii) A diagnosis of a familial or hereditary condition known to be associated with phaeochromocytoma (multiple endocrine neoplasia, von Hippel-Landau disease, neurofibromatosis, etc).

   All subjects: (enrolled under Amendments 01 and 02)
2. The subject is able and willing to comply with study procedures and a signed and dated informed consent is obtained.
3. The subject was male; or a female who was either pre-menarchal, surgically sterile (had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test (with the results known prior to investigational medicinal product (IMP) administration) was negative.

Exclusion Criteria:

1. The subject was previously entered into this study or had participated in any other investigational medicinal product or medical device study within 30 days of enrolment.
2. The subject had a history or suspicion of significant allergic reaction or anaphylaxis to iodide or iodinated imaging agents.
3. The subject presented with any clinically active, serious, life-threatening disease other than neuroblastoma or phaeochromocytoma, with a life expectancy of less than 30 days or where participation in the study would compromise the management of the subject or other reason that in the judgement of the investigator(s) made the subject unsuitable for participation in the study.
4. The subject had a history of renal insufficiency (serum creatinine >3.0 mg/dL [265 μmol/L]).
5. The subject used medications that are known to interfere with 123I-mIBG uptake and these medications could not be safely withheld for at least 24 hours before study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2005-08-02 (Actual); Primary Completion 2006-09-27 (Actual); Study Completion 2006-09-27 (Actual)

PRIMARY OUTCOMES:
- To demonstrate that 123I-mIBG planar scintigraphy is sensitive and specific in confirming or excluding the diagnoses of neuroblastoma and phaeochromocytoma.

SECONDARY OUTCOMES:
To determine the incremental value of single-photon emission computed tomography (SPECT) for improving the sensitivity and specificity of 123I-mIBG planar scintigraphy for the diagnoses of neuroblastoma and phaeochromocytoma.
To collect safety data on 123I-mIBG.

CONTACTS AND LOCATIONS:
Overall Officials: Diane McCaul, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States